CLINICAL TRIAL: NCT00986362
Title: The MIC (Microplasmin In Children) Trial: A Randomized, Placebo-controlled, Double-masked, Clinical Trial of Intravitreal Microplasmin in Infants and Children Scheduled for Vitrectomy
Brief Title: Clinical Trial of Intravitreal Microplasmin in Infants and Children Scheduled for Vitrectomy
Acronym: MIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-MV-009
Record Dates: First submitted 2009-09-28; First posted 2009-09-29 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Vitrectomy
Keywords: Safety in pediatrics
MeSH Terms: interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ocriplasmin (Experimental)
  Interventions: Drug: Ocriplasmin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocriplasmin — 175µg ocriplasmin intravitreal injection
  Arms: Ocriplasmin
Drug: Placebo — Placebo intravitreal injection
  Arms: Placebo

SUMMARY:
To evaluate the safety and preliminary efficacy of intravitreal microplasmin as an adjunct to conventional vitrectomy for the treatment of pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants or children 16 years of age or younger
2. Patient must be a suitable candidate for conventional 2-port or 3-port pars plana vitrectomy
3. Patient with attached vitreous somewhere in posterior pole
4. Patient's parent or guardian must be willing and able to comply with follow-up requirements
5. Patient's parent(s) must sign informed parental permission form and in the case of school-age children the patient must sign assent form

Exclusion Criteria:

1. Patient diagnosed with Stage 1, 2, 3 or 5 retinopathy of prematurity (ROP) at the time of surgery
2. Unclear media, which precludes assessment of the posterior pole such as a cataract or vitreal opacity
3. Active parental/guardian drug or alcohol use or dependence that, in the opinion of the site Investigator, would interfere with parent's or guardian's adherence to study requirements
4. Medical problems that make consistent follow-up over the treatment period uncertain.
5. Patient must not have participated in an investigational drug or device study in the prior 30 days
6. Female Patients of childbearing potential must not be pregnant or lactating.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Associated Retina Consultants, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was recruited on 10 Feb 2010 and last subject completed the study on 14 Dec 2011.
  24 study eyes (16 ocriplasmin, 8 placebo) were evaluated during the study. 22 subjects were enrolled in the study. 2 subjects were treated in both eyes.
Groups:
- Ocriplasmin: Ocriplasmin : 175µg ocriplasmin intravitreal injection
- Placebo: Placebo : Placebo intravitreal injection
Period: Overall Study
Arm/Group | Ocriplasmin | Placebo
Started | 16 (16 eyes randomized and treated (in 15 subjects).) | 8 (8 eyes randomized and treated (in 8 subjects).)
Completed | 14 (14 eyes completed the study (in 14 subjects).) | 7 (7 eyes completed the study (in 7 subjects).)
Not Completed | 2 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 16 eyes randomized and treated (in 15 subjects) with ocriplasmin & 8 eyes randomized and treated (in 8 subjects) with placebo. Randomisation was at the eye not the subject level; in 1 subject, both eyes were randomised to ocriplasmin; in 1 subject, 1 eye was randomised to ocriplasmin & 1 eye randomised to placebo. 22 subjects participated, 24 eyes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (6.40) | 8.0 (6.61) | 6.8 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Total Macular Posterior Vitreous Detachment (PVD).
Description: Percentage of eyes with total macular PVD (to the vascular ridge in eyes with ROP) at the beginning of vitrectomy or after application of suction, as assessed by masked surgeon observation under the operating microscope.
Time Frame: Beginning of vitrectomy or after application of suction
Population: Study eyes were analysed according to the Intent-to-Treat (ITT) principle, i.e. as randomised regardless of treatment received. The primary endpoint was evaluated using the Full Analysis Set (FAS), with missing data imputed using the Last Observation Carried Forward (LOCF) method. 1 subject contributed 1 eye to both treatment groups
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Ocriplasmin | Placebo
Number analyzed (Participants) | 15 | 8
Number analyzed (Eyes) | 16 | 8
percentage of eyes | 50 | 62.5
Statistical Analysis 1: Comparison: Ocriplasmin vs Placebo; Test type: Superiority or Other; p = 0.679, Fisher Exact; Odds Ratio (OR) = 0.613, 95% CI 2-sided [0.070 to 4.509]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs)/Serious Adverse Events (SAEs) were collected from the study drug administration day to the end of study (6 months follow-up visit).
Description: The reporting for the study was made based in number of eyes and not in the number of participants, therefore the number of "participants" at risk in the AE section is actually the number of "eyes" at risk.
Arm/Group | Ocriplasmin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/16 | 2/8
Other Adverse Events (participants affected / at risk) | 15/16 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin (N=16) | Placebo (N=8)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin (N=16) | Placebo (N=8)
Eye pain (Eye disorders) | 12 (12) | 4 (4)
Eyelid oedema (Eye disorders) | 6 (6) | 5 (5)
Conjunctival haemorrhage (Eye disorders) | 7 (7) | 4 (4)
Anterior chamber cell (Eye disorders) | 5 (5) | 3 (3)
Anterior chamber flare (Eye disorders) | 5 (7) | 3 (4)
Conjunctival hyperaemia (Eye disorders) | 3 (3) | 3 (3)
Maculopathy (Eye disorders) | 6 (10) | 3 (5)
Corneal epithelium defect (Eye disorders) | 1 (1) | 2 (2)
Retinal detachment (Eye disorders) | 4 (5) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 4 (4) | 1 (1)
Retinal disorder (Eye disorders) | 3 (3) | 0 (0)
Blepharospasm (Eye disorders) | 2 (2) | 0 (0)
Chorioretinal disorder (Eye disorders) | 0 (0) | 1 (1)
Chromatopsia (Eye disorders) | 0 (0) | 1 (1)
Conjunctival oedema (Eye disorders) | 2 (2) | 1 (1)
Corneal disorder (Eye disorders) | 1 (1) | 1 (1)
Corneal oedema (Eye disorders) | 1 (1) | 1 (1)
Corneal thickening (Eye disorders) | 0 (0) | 1 (1)
Cyclitic membrane (Eye disorders) | 2 (2) | 0 (0)
Glaucomatous optic disc atrophy (Eye disorders) | 0 (0) | 1 (1)
Hypotony of eye (Eye disorders) | 2 (3) | 0 (0)
Macular oedema (Eye disorders) | 2 (2) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1) | 1 (1)
Optic atrophy (Eye disorders) | 2 (2) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Retinal oedema (Eye disorders) | 2 (3) | 1 (2)
Retinal pigment epitheliopathy (Eye disorders) | 2 (2) | 1 (1)
Retinal tear (Eye disorders) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Anterior chamber fibrin (Eye disorders) | 1 (2) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Ciliary zonular dehiscence (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Corneal opacity (Eye disorders) | 1 (2) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0)
Hyphaema (Eye disorders) | 1 (3) | 0 (0)
Iris adhesions (Eye disorders) | 1 (1) | 0 (0)
Iris bombe (Eye disorders) | 1 (1) | 0 (0)
Iris neovascularization (Eye disorders) | 1 (1) | 0 (0)
Lacrimal haemorrahge (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Optic nerve sheath haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Pupillary disorder (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0)
Subretinal fibrosis (Eye disorders) | 1 (1) | 0 (0)
Vitreous adhesions (Eye disorders) | 1 (1) | 0 (0)
Vitreous disorder (Eye disorders) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Shunt infection (Infections and infestations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 3 (3)
Foreign body in eye (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Optic nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Retinal scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Device malfunction (General disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less